CLINICAL TRIAL: NCT02479256
Title: Clomiphene Citrate Versus Tamoxifen for Induction of Ovulation in Women With Polycystic Ovary Syndrome: Randomized Controlled Trial
Brief Title: Clomiphene Citrate Versus Tamoxifen for Ovulation Induction in PCOs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20092009
Record Dates: First submitted 2015-04-13; First posted 2015-06-24 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: PCOS
Keywords: PCOS; Induction of ovulation; Clomiphene citrate; Tamoxifen
MeSH Terms: interventions — Clomiphene; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomiphene citrate + placebo (Experimental): Women will receive one tablet of clomiphene citrate oral tablets 50 mg (Clomid®, aventis/Egypt) twice daily 12 hours apart (total dose 100 mg daily), and one tablet of placebo of tamoxifen oral tablets twice daily 12 hours apart from the 3rd day of the menses for 5 days, for only one menstrual cycle.
  Interventions: Drug: Clomiphene citrate; Drug: Tamoxifen Placebo
- Tamoxifen + placebo (Experimental): Women will receive one tablet of tamoxifen oral tablets 10 mg (Tamoxifen®, amriya/Egypt) twice daily 12 hours apart (total dose 20 mg daily), and one tablet of placebo of clomiphene citrate twice daily 12 hours apart from 3rd day of the menses for 5 days, for only one menstrual cycle.
  Interventions: Drug: Tamoxifen; Drug: Clomiphene citrate placebo

INTERVENTIONS:
Drug: Clomiphene citrate — Women will receive one tablet of clomiphene citrate oral tablets 50 mg (Clomid®, aventis/Egypt) twice daily 12 hours apart (total dose 100 mg daily) from the 3rd day of the menses for 5 days, for only one menstrual cycle.
  Other Names: Clomid
  Arms: Clomiphene citrate + placebo
Drug: Tamoxifen Placebo — Women will receive one tablet of placebo of tamoxifen oral tablets twice daily 12 hours apart from the 3rd day of the menses for 5 days, for only one menstrual cycle.
  Arms: Clomiphene citrate + placebo
Drug: Tamoxifen — Women will receive one tablet of tamoxifen oral tablets 10 mg (Tamoxifen®, amriya/Egypt) twice daily 12 hours apart (total dose 20 mg daily) from 3rd day of the menses for 5 days, for only one menstrual cycle.
  Arms: Tamoxifen + placebo
Drug: Clomiphene citrate placebo — Women will receive one tablet of placebo of clomiphene citrate twice daily 12 hours apart from 3rd day of the menses for 5 days, for only one menstrual cycle.
  Arms: Tamoxifen + placebo

SUMMARY:
Comparison between Clomiphene citrate and Tamoxifen for induction of ovulation in women with PCOS.

DETAILED DESCRIPTION:
Participants fulfilling inclusion and exclusion criteria will be divided into two groups, each group containing 300 participants;

Group (A):

300 participants will receive Clomiphene citrate oral tablets and placebo of Tamoxifen oral tablets.

Group (B):

300 participants will receive Tamoxifen oral tablets and placebo of Clomiphene oral tablets.

Participants with abnormal menstrual history will receive two tablets of norethisterone 5mg tab (Steronate nor ®, hi pharm/Egypt) every12 hours for 5 days to withdraw period before starting the procedure.

Then;

Group (A):

Women will receive one tablet of clomiphene citrate oral tablets 50 mg (Clomid®, aventis/Egypt) twice daily 12 hours apart (total dose 100 mg daily), and one tablet of placebo of tamoxifen oral tablets twice daily 12 hours apart from the 3rd day of the menses for 5 days, for only one menstrual cycle.

Group (B):

Women will receive one tablet of tamoxifen oral tablets 10 mg (Tamoxifen®, amriya/Egypt) twice daily 12 hours apart (total dose 20 mg daily), and one tablet of placebo of clomiphene citrate twice daily 12 hours apart from 3rd day of the menses for 5 days, for only one menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Primary infertility.
* Body mass index (BMI) between 25 and 30 Kg/m 2.
* Polycystic ovary syndrome (using ESHRE/ASRM criteria).

Exclusion Criteria:

* Secondary infertility.
* Patients with BMI under 25 or over 30 Kg/m 2.
* Hyper or hypothyroidism, or hyperprolactinemia.
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugs.
* Intention to start a diet or a specific program of physical activity.
* Organic pelvic diseases.
* Tubal or male factor infertility.
* Interval of earlier treatment with any of the fertility drugs of less than 6 months.
* Contraindication to either:

  * Clomiphene citrate.
  * Tamoxifen.
  * HCG injection.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of ovulation. | Up to 4 weeks from starting treatment.
  * Transvaginal ultrasound done to:
    1. Detect signs of ovulation: corpus luteum, fluid in cul-de-sac, collapse of the follicle size.
  * Serum progesterone will be measured in the mid luteal day of the cycle, where:
    1. Level 6 ng/ml or 19 nmol/L indicates Ovulation.
    2. Level <5 nmol/L suggests Ovulation did not occur.

SECONDARY OUTCOMES:
Endometrial perfusion by using 3D- power Doppler (GE Medical system volouson E6, 5-7 MHz) in the mid luteal day of the cycle to assess endometrial receptivity. | Up to 4 weeks from starting treatment.
  Endometrial perfusion by using 3D-power Doppler (GE Medical system volouson E6, 5-7 MHz) at Ain-Shams University Maternity Hospital will be done in the mid luteal day of the menstrual cycle to assess endometrial receptivity by measured:
  * Gray: mean Gray value.
  * Color angio: Flow index, Vascularization index, and Vascularization flow Index.
Endometrial thickness and quality in the pre-ovulatory period. | Up to 4 weeks from starting treatment.
  Transvaginal ultrasound will be done to:
  Evaluate endometrial thickness and quality pre-ovulatory: where the minimal endometrial thickness to achieve a pregnancy ranges from 4 to 7mm with a healthy trilaminar appearance.
Number of growing follicles detected by transvaginal ultrasound. | Up to 4 weeks from starting treatment.
  Transvaginal ultrasound will be done to:
  Detect mean follicular diameter in the days 10, 12, 14 and up to day 25 of the cycle.
Pregnancy rate both clinical and biochemical. | Up to 8 weeks from starting treatment.
  Transvaginal ultrasound done to:
  1. Evaluate endometrial thickness and quality in the mid luteal day of the cycle: where the optimal endometrial thickness to achieve a pregnancy ranging from 10 to 15mm with a healthy trilaminar appearance.
  2. Detect gestational and fetal pulsation.
Patient compliance. | Up to 4 weeks from starting treatment.
  Asking the participant about the empty strips.
Adverse effects: such as headache, nausea, vomiting, breast tenderness, blurred vision, and ovarian enlargement or hyperstimulation. | Up to 4 weeks from starting treatment.
  Asking the participant if there are any complaints about the side effects of the drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Gasser M. El-Bishry, FRCOG, Study Director — Professor of Obstetrics and Gynaecology, Ain Shams University; Abdel-Latif G. El-Kholy, MD, Principal Investigator — Assistant professor of Obstetrics and Gynaecology, Ain Shams University; Mohamed S. Sweed, MD, Principal Investigator — Lecturer of Obstetrics and Gynaecology, Ain Shams University; Diana N. Kolta, MB BCh, Principal Investigator — Resident of Obstetrics and Gynaecology
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt